CLINICAL TRIAL: NCT06780176
Title: Genomic and Non-Genomic Factors Associated With Breast Cancer Risk Factors and Outcomes in a Diverse South Florida Population
Brief Title: A Study of Breast Cancer Risk Factors and Outcomes of People in Florida
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-372
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Diseases
Keywords: breast cancer; breast neoplasms; breast diseases; BIRADS; Memorial Sloan Kettering Cancer Center; 24-372
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional blood and/or tissue samples at the time of participant scheduled biopsy procedure in radiology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with BIRADS 0-5: Men and woman 18 years and older who are participants with BIRADS 0-5 who present to breast radiology for biopsy or any new breast patient.
  Interventions: Other: Biospecimen Collection; Diagnostic Test: Surgical Tissue Collection; Behavioral: Survey Collection

INTERVENTIONS:
Other: Biospecimen Collection — Blood collection at baseline and time of surgery
Diagnostic Test: Surgical Tissue Collection — Tissue collection will be attempted at time of surgery
Behavioral: Survey Collection — Survey collection at baseline, post-surgery, at 1, 3 and 5 year follow up visits

SUMMARY:
The purpose of this study is to understand why different people have different risks and outcomes for breast cancer and non-breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BIRADS 0-5, seen in breast radiology clinic at University of Miami (UM), Sylvester Comprehensive Cancer Center (SCCC), Jackson Health Systems (JHS) for biopsy.
* Any new breast patient seen at UM/SCCC or JHS will be invited to participate in the study.
* Men and women 18 years of age and older are eligible to participate in the study.

Exclusion Criteria:

* Patients who are less than 18 years of age will be considered ineligible.
* Patients unable to complete the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Miami treating clinicians will identify participants (anyone meeting inclusion criteria listed above) during their regularly scheduled visits (Breast radiology at time of initial biopsy, Surgery clinic visit, Medical Oncology clinic visit) or in the pre-operative waiting area prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2030-01-13 (Estimated); Study Completion 2030-01-13 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristic of participants (survey) | Up to 5 years
  The purpose of this study is to prospectively collect and store clinical data, blood and tissue samples, and participant survey data to evaluate (epi) genomic and non-genomic causes of disparity.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Goel, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - University of California, Los Angeles (Specimen Analysis only), Los Angeles, California
  - University of Miami (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org